CLINICAL TRIAL: NCT04071665
Title: A Modified Lateral Lumbar Interbody Fusion VS. Transforaminal Lumbar Interbody Fusion for Adult Degenerative Scoliosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); First Affiliated Hospital of Shantou University Medical College (Other); Shenzhen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSFC 81702220
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2019-06

CONDITIONS: Degenerative Scoliosis; Minimally Invasive; Spinal Deformity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified lateral lumbar interbody fusion (Experimental): Modified lateral lumbar interbody fusion for treatment of scoliosis
  Interventions: Procedure: Modified lateral lumbar interbody fusion
- transforaminal lumbar interbody fusion (Active Comparator): transforaminal lumbar interbody fusion
  Interventions: Procedure: Modified lateral lumbar interbody fusion

INTERVENTIONS:
Procedure: Modified lateral lumbar interbody fusion — Modified lateral lumbar interbody fusion

SUMMARY:
A modified lateral lumbar interbody fusion VS. transforaminal lumbar interbody fusion for the treatment of adult degenerative scoliosis with 2 year follow-up with a multiple center, randomized case-control study

DETAILED DESCRIPTION:
Adult degenerative scoliosis (ADS) is the most common spinal deformity in the elderly, and the severe patients need surgical treatment. The elderly are often complicated with many medical diseases and the perioperative risk is high, so minimally invasive surgery is a new choice for spinal surgeons to treat ADS. Modified lateral lumbar interbody fusion (CLIF) is an new modified spinal minimally invasive interbody fusion technique in the investigator's department. The results of preliminary studies showed that it has the advantages of less trauma, short operation time and fewer complications, and the clinical and imaging outcome are remarkable. Therefore, the present study aims to establish a multicenter, large sample prospective randomized controlled study to explore the technical advantages and surgical indications of the new technique in the treatment of ADS by comparing with the traditional posterior spinal interbody fusion; (2) to compare the postoperative clinical and imaging results and analyze the surgical complications and preventive measures; (3) to establish a long-term follow-up to further quantify the clinical and imaging outcome of the new technique. Therefore, this study will further verify the safety and effectiveness of the CLIF in the treatment of ADS on the basis of previous studies, and provide a new clinical approach for minimally invasive treatment of ADS.

ELIGIBILITY:
Inclusion Criteria:

* at least 50 years of age, diagnosed with adult thoracolumbar scoliosis including any number of intervertebral levels between T8 and S1, unresponsive to conservative treatment for at least 6 months, and had a preoperative coronal Cobb angle of at least 10° and preoperative ODI score of at least 30%.

Exclusion Criteria:

* with prior lumbar fusion surgery or spondylolisthesis greater than Grade II

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
ODI score | 2 years
  an index for assessing the lower back pain wiith multiple questionnare

CONTACTS AND LOCATIONS:
Overall Officials: Qixin CHEN, Ph.D, Study Director — Orthopedics Department, 2nd Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
after complete the recruiment with half of participants, we will share the preliminary results with data.

REFERENCES:
- [Background] Mendoza-Lattes S. Cervical Disc Replacement: Are We There Yet? Commentary on an article by Michael E. Janssen, DO, et al.: "ProDisc-C Total Disc Replacement Versus Anterior Cervical Discectomy and Fusion for Single-Level Symptomatic Cervical Disc Disease. Seven-Year Follow-up of the Prospective Randomized U.S. Food and Drug Administration Investigational Device Exemption Study". J Bone Joint Surg Am. 2015 Nov 4;97(21):e71. doi: 10.2106/JBJS.O.00750. No abstract available. PMID 26537171
- [Background] Kretzer RM. Adult Degenerative Spinal Deformity: Overview and Open Approaches for Treatment. Spine (Phila Pa 1976). 2017 Apr 1;42 Suppl 7:S16. doi: 10.1097/BRS.0000000000002028. No abstract available. PMID 28296697
- [Background] Bach K, Ahmadian A, Deukmedjian A, Uribe JS. Minimally invasive surgical techniques in adult degenerative spinal deformity: a systematic review. Clin Orthop Relat Res. 2014 Jun;472(6):1749-61. doi: 10.1007/s11999-013-3441-5. PMID 24488750
- [Result] Epstein NE. Commentary on: Laminectomy plus fusion versus laminectomy alone for lumbar spondylolisthesis by Ghogawala Z, Dziura J, Butler WE, Dai F, Terrin N, Magge SN, et al. NEJM 2016;374 (15):1424-34. Surg Neurol Int. 2016 Sep 22;7(Suppl 25):S644-S647. doi: 10.4103/2152-7806.191061. eCollection 2016. PMID 27843677
- [Result] Epstein NE. Commentary on: A randomized controlled trial of fusion surgery for lumbar spinal stenosis (Forsth P, Olafsson G, Carlsson T, Frost A, Borgstrom F, Fritzell P, et al. N Eng J Med 2016;374:1414-23). Surg Neurol Int. 2016 Sep 22;7(Suppl 25):S641-S643. doi: 10.4103/2152-7806.191060. eCollection 2016. PMID 27843676